CLINICAL TRIAL: NCT06593340
Title: Evaluation of Report-Back Strategies for Long-term and Short-term Exposure Information in Rural Tribal Populations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Darrah Sleeth, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01ES036260 (NIH); R01ES036260 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Behavior Change
Keywords: exposure; Native American; radon; particulate matter; PM2.5; report-back
MeSH Terms: interventions — IGF2BP3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-Time Exposure Data (Experimental): Participants in this arm will get their data reported-back in real-time. There will be a total of 4 different strategies tested based on a combination of two (2) messengers and two (2) formats tested.
  Interventions: Behavioral: Messenger 1; Behavioral: Messenger 2; Behavioral: Format 1; Behavioral: Format 2
- Delayed Exposure Data (Experimental): Participants in this arm will get their data reported-back only after all exposure data are collected (i.e., delayed approximately 2 months). There will be a total of 4 different strategies tested based on a combination of two (2) messengers and two (2) formats tested.
  Interventions: Behavioral: Messenger 1; Behavioral: Messenger 2; Behavioral: Format 1; Behavioral: Format 2

INTERVENTIONS:
Behavioral: Messenger 1 — The first type of messenger (specific details TBD) that will be used to deliver the environmental sampling results.
Behavioral: Messenger 2 — The second type of messenger (specific details TBD) that will be used to deliver the environmental sampling results.
Behavioral: Format 1 — The first type of format (specific details TBD) that will be used to deliver the environmental sampling results.
Behavioral: Format 2 — The second type of format (specific details TBD) that will be used to deliver the environmental sampling results.

SUMMARY:
The goal of this study is to evaluate different ways to provide feedback about environmental sampling results to participants. Specifically, the study will look at exposures with long-term risk (radon) and short-term risk (indoor particulate matter, PM2.5). The hypothesis is that providing feedback in real-time will result in participants engaging in more activities to try to reduce their exposure. One of the main questions of interest is: How does the information messenger impact the effectiveness of report-back strategies in rural, tribal populations?

Participants will have radon and PM2.5 measurement equipment installed at their home and will answer questions about any actions they took to reduce exposure. Previously developed approaches to reporting back those exposures will be used to test which feedback method results in more actions to reduce exposure.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled member of the participating tribe

Exclusion Criteria:

* Participant in one of our previous studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Exposure Reduction Behaviors | 3 months after report-back
  This will be collected using a questionnaire with a likert scale from 1 (not at all) to 10 (a lot) of how often certain exposure-reduction behaviors are performed.
Exposure Reduction Behaviors | 6 months after report-back
  This will be collected using a questionnaire with a likert scale from 1 (not at all) to 10 (a lot) of how often certain exposure-reduction behaviors are performed.
Exposure Reduction Behaviors | 12 months after report-back
  This will be collected using a questionnaire with a likert scale from 1 (not at all) to 10 (a lot) of how often certain exposure-reduction behaviors are performed.

IPD SHARING:
Plan to Share IPD: No